CLINICAL TRIAL: NCT01983696
Title: The Effect of Low Oxygen Tension on the Early Development of Human Embryo in IVF/ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Provincial Maternity and Children's Hospital (Other)
Responsible Party: Principal Investigator, Shi Wenhao, Assisted Reproductive Technology Center, Shanxi Provincial Maternity and Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCHC-2013-02
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Embryo Hypoxia
Keywords: low oxygen tension; embryo quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5% oxygen (Experimental): the oocytes and embryos are cultured in 5% oxygen concentration after oocytes retrieval until Day 6 (counting from fertilization)
  Interventions: Other: 5% oxygen concentration
- 20% oxygen (No Intervention): the oocytes and embryos are cultured in 20% oxygen concentration (in atmosphere) after oocytes retrieval until Day 6(counting from fertilization)

INTERVENTIONS:
Other: 5% oxygen concentration — the oocytes and embryos are cultured in the incubator with concentrations of 6% CO2,5%O2, and 89% N2
  Other Names: low oxygen concentration
  Arms: 5% oxygen

SUMMARY:
To investigate the effect of low oxygen tension during in vitro culture in terms of embryo quality and outcomes of pregnancy in vitro fertilization/ Intracytoplasmic sperm injection

DETAILED DESCRIPTION:
The oocytes will be divided into two parts(two groups) form one patient. The two groups of oocytes will be cultured seperately in the incubator with the concentrations of 5% CO2,6%O2,89% N2(low oxygen concentration) verse 6% CO2,20% O2,74% N2(in atmosphere).

A series of observational measurement(embryo quality and outcomes of pregnancy) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Fresh cycles of in vitro fertilization/intracytoplasmic sperm injection and emrbyo transfer (IVF/ICSI-ET)
* ≥ 10 oocytes after oocyte retrieval

Exclusion Criteria:

* ≥ 3 transfer or oocyte retrieval cycles
* PGD/PGS cycles
* half-ICSI/rescure ICSI
* fluid in the uterine cavity, abnormal endometrium, uterine abnormalities,pelvic inflammation
* acute maternal problems.
* One or both spouses have an abnormal karyotype (including polymorphism)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
embryo quality | up to 6 days after fertilization
  Embryo morphology was assessed on day 2, day 3 day 4 day 5 day and 6 by considering the number of blastomeres, symmetry and granularity of blastomeres, type and percentage of fragmentation, presence of multinucleated blastomeres, and degree of compaction.
  Gardner's blastocyst scoring system is used for blastocyst assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Shi, Master, Study Director — Maternal and Children Health Care Hospital
Locations (1):
- Maternal and Child Health Care Hospital, Xi'an, Shaanxi, China